CLINICAL TRIAL: NCT05458193
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Crossover Study to Investigate the Effects of Daridorexant on Nighttime Respiratory Function and Sleep in Patients With Severe Obstructive Sleep Apnea
Brief Title: A Study to Investigate the Effects of Daridorexant on Nighttime Breathing in Patients With Shallow or Paused Breath During Sleep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-078-121; 2022-000098-23 (EudraCT Number)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Obstructive Sleep Apnea of Adult
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: 2-way cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daridorexant (Experimental): 50 mg once daily from Day 1 to Day 5
  Interventions: Drug: Daridorexant
- Placebo (Placebo Comparator): Matching placebo once daily from Day 1 to Day 5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant — Film-coated tablet for oral use
  Other Names: ACT-541468
  Arms: Daridorexant
Drug: Placebo — Film-coated tablet for oral use
  Arms: Placebo

SUMMARY:
A study on the effects of daridorexant on nighttime respiratory function in patients with severe obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Each subject will participate in 2 study periods. Participants will receive 50 mg daridorexant in one period and placebo in the other period. Both periods will last from Day 1 (first administration) in the evening to Day 6 in the morning (defined as End-of-Period). The 2 periods will be separated by an in-between period of 1 to 2 weeks. An End-of-Study examination will take place 1 to 2 weeks after last administration of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Male and female participants aged 18 years or older at Screening.
* Diagnosis of Obstructive Sleep Apnea (OSA) according to the International Classification of Sleep Disorders, documented by medical history and confirmed by a specialist.
* Severe intensity of OSA determined during OSA diagnosis and confirmed during both screening night polysomnography (PSG) and defined as apnea/hypopnea index greater than or equal to 30 events per hour.
* Patient who may require a continuous positive airway pressure (CPAP) device or a dental appliance device for the treatment of OSA must either not have started it or have withdrawn from it at least 2 months before randomization in this study. In all cases patients must not start using this type of device during the study.
* Women of childbearing potential must have a negative serum pregnancy test at Screening Visit 1 and a negative urine pregnancy test on Day 1 pre-dose of the first study period. She must agree to consistently and correctly use a highly effective method of contraception with a failure rate of less than 1% per year, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must be initiated at least 1 month before first treatment administration.
* Woman of non-childbearing potential, i.e., postmenopausal, with previous bilateral salpingectomy, bilateral salpingo-oophorectomy or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, or uterine agenesis.

Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity or vulnerability (e.g., kept in detention) at Screening.
* Pregnant or lactating woman.
* Modified Swiss Narcolepsy Scale total score less than 0 at Screening or history of narcolepsy or cataplexy.
* Participant with clinically significant abnormality present on either or both screening night PSG.
* Evidence of any other clinically significant active pulmonary disease such as chronic obstructive pulmonary disease (as per Global Initiative for Obstructive Lung Disease), based on investigator's judgment.
* History of surgical intervention for OSA, except nose surgery.
* Subject is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff from study site or the sponsor directly involved in the conduct of the study or their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Treatment difference (daridorexant - placebo) for apnea/hypopnea index | Night 5 of period 1 and period 2 (Total duration: 2 days)
  The treatment difference will be assessed at Night 5 of period 1 and period 2 after repeated-dose administration, as measured by polysomnography.
  Polysomnography recording will start at the time of "lights off" and last for 8 hours.
  The apnea/hypopnea index is defined by the total number of apneas (pause in respiration ≥ 10 sec) plus hypopneas (peak signal excursions drop by ≥ 30% of pre-event baseline for at least 10 sec accompanied by a decrease of SpO2 ≥ 3% from pre-event baseline and/or the event is associated with an arousal) during total sleep time (TST), divided by TST (in min), then multiplied by 60.

SECONDARY OUTCOMES:
Treatment difference (daridorexant - placebo) in mean peripheral oxygen saturation (SpO2) during total sleep time | Night 5 of period 1 and period 2 (Total duration: 2 days)
  The treatment difference will be assessed at Night 5 of period 1 and period 2 after repeated-dose administration, as measured by pulse oximetry.
  Pulse oximetry recording will start at the time of "lights off" and last for 8 hours.
Treatment difference (daridorexant - placebo) for total sleep time | Night 5 of period 1 and period 2 (Total duration: 2 days)
  The treatment difference will be assessed at Night 5 of period 1 and period 2 after repeated-dose administration, as measured by polysomnography.
  Polysomnography recording will start at the time of "lights off" and last for 8 hours.
Daridorexant plasma concentration | 9 hours post-dose on Day 2 and Day 6 (Total duration: up to 2 days)
Incidence of treatment-emergent adverse events | Day 1 up to Day 13 (Total duration: 13 days)
  A treatment-emergent adverse event is any adverse event temporally associated with the use of a study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- ASR Advanced Sleep Research GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No